CLINICAL TRIAL: NCT03394781
Title: A Randomized, Open-label, Phase 2 Study to Evaluate Safety and Efficacy of DUR-928 in Subjects With Primary Sclerosing Cholangitis (PSC)
Brief Title: A Research Study to Evaluate Safety and Efficacy of DUR-928 in Subjects With Primary Sclerosing Cholangitis (PSC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Durect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C928-008
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-08

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DUR-928 10 mg (Experimental): 10 mg oral suspension
  Interventions: Drug: DUR-928
- DUR-928 50 mg (Experimental): 50 mg oral suspension
  Interventions: Drug: DUR-928

INTERVENTIONS:
Drug: DUR-928 — oral suspension daily for 28 days

SUMMARY:
This is a research trial testing DUR-928 (an experimental medication). The purpose of the trial is to assess whether treatment with DUR-928 has any effect on the treatment of Primary Sclerosing Cholangitis (PSC). This trial will also assess safety (side effects).

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of primary sclerosing cholangitis (PSC) for at least 12 months, with or without inflammatory bowel disease (IBD).
* Serum alkaline phosphatase (ALP) ≥ 1.5 times ULN and with no >15% fluctuation in the past 3 months.
* In subjects receiving treatment with ursodeoxycholic acid (UDCA), therapy must be stable for at least 3 months and at a dose not greater than 20 mg/kg/day.
* Subjects of childbearing potential must agree to use a medically acceptable method of contraceptive to prevent pregnancy in the subject and/or the partner for the duration of their participation in the trial up to 2 months after the last study drug dosing.

Exclusion Criteria:

* Presence of documented secondary sclerosing cholangitis or small duct PSC
* Bacterial cholangitis within 30 days prior to Screening
* Presence of percutaneous drain or endoscopic bile duct stent
* History of, or suspicion of cholangiocarcinoma.
* Prior liver transplantation, or currently listed for liver transplantation
* Presence of other concomitant liver diseases
* Moderate to Severe active IBD or flare in colitis activity within the last 3 months
* Any severe and/or untreated concomitant cardiovascular, renal, endocrine or psychiatric disorder
* Any active malignant disease (within 3 years), other than non-melanomatous skin cancer
* Human immunodeficiency virus (HIV) infection
* Existing or intended pregnancy, or breast feeding
* Has received medication from another clinical trial within the past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Smith, MD, Study Director — INC Research/InVentiv Health
Locations (4):
- United States (4):
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Charlotte Mecklenburg Hospital, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated early due to lack of enrollment.
Period: Overall Study
Arm/Group | DUR-928 10 mg | DUR-928 50 mg
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DUR-928 10 mg | DUR-928 50 mg | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Alkaline Phosphatase (ALP) From Baseline
Time Frame: Day 28 (end of treatment) and Day 56 (end of study/early termination)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DUR-928 10 mg | DUR-928 50 mg
Number analyzed (Participants) | 3 | 2
percent change
  Percent change of ALP from baseline to Day 28 | 23.7 (10.7) | 16.8 (2.97)
  Percent change of ALP from baseline to Day 56 | 10.7 (17.04) | 11.05 (8.68)

2. Secondary Outcome: Percent Change of Liver Enzymes and Serum Bile Acids (sBA)
Description: Liver enzymes include alanine transaminase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), bilirubin.
  Percent change from baseline through the end of study treatment (Day 28) and throughout the follow-up period (Day 56).
Time Frame: Day 28 and Day 56
Population: Study terminated early due to lack of enrollment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DUR-928 10 mg | DUR-928 50 mg
Number analyzed (Participants) | 3 | 2
percent change
  percent ALT change from baseline to Day 28 | 32.87 (48.87) | 3.0 (29.56)
  percent AST change from baseline to Day 28 | 24.10 (35.03) | -20.25 (3.23)
  percent GGT change from baseline to Day 28 | 7.3 (4.16) | 8.15 (1.49)
  percent direct bilirubin change from baseline to Day 28: number analyzed (Participants) | 2 | 1
  percent direct bilirubin change from baseline to Day 28 | 14.2 (24.61) | 34.6 (NA) — Standard Deviation not calculable because data were only collected for 1 participant.
  percent total bilirubin change from baseline to Day 28 | 12.03 (23.09) | 23.85 (33.73)
  percent serum bile acids change from baseline to Day 28 | -13.93 (15.00) | -44.10 (46.95)
  percent ALT change from baseline to Day 56 | -9.77 (15.30) | -12.7 (5.66)
  percent AST change from baseline to Day 56 | -16.23 (9.17) | -9.70 (19.09)
  percent GGT change from baseline to Day 56 | -7.10 (11.87) | -3.2 (2.26)
  percent direct bilirubin change from baseline to Day 56: number analyzed (Participants) | 1 | 1
  percent direct bilirubin change from baseline to Day 56 | -12.90 (NA) — Standard Deviation not calculable because data were only collected for 1 participant. | 19.20 (NA) — Standard Deviation not calculable because data were only collected for 1 participant.
  percent total bilirubin change from baseline to Day 56 | -24.60 (20.46) | 19.14 (15.61)
  percent serum bile acids change from baseline to Day 56 | 35.23 (79.79) | -35.75 (72.90)

3. Secondary Outcome: Percent of Subjects With Reduction of Serum Alkaline Phosphatase (ALP) From Baseline
Time Frame: Day 28 (end of treatment) and Day 56 (end of follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | DUR-928 10 mg | DUR-928 50 mg
Number analyzed (Participants) | 3 | 2
Participants
  subjects with ≥ 40% reduction of serum ALP from baseline at day 28/end of treatment | 0 | 0
  subjects with ≥ 40% reduction of serum ALP from baseline at day 56/end of follow-up | 0 | 0

4. Secondary Outcome: Percent Change of Selected Biomarkers From Baseline Through the End of Study Treatment and Throughout the Follow-up Period.
Time Frame: Day 28 and Day 56
Population: The samples were not assayed to generate data for this Outcome Measure due to early study termination.
Arm/Group | DUR-928 10 mg | DUR-928 50 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 days
Description: Treatment Emergent Adverse Events
Arm/Group | DUR-928 10 mg | DUR-928 50 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DUR-928 10 mg (N=3) | DUR-928 50 mg (N=2)
DRUG INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
WORSENING SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
EXCESSIVE GAS (FLATUS) (Gastrointestinal disorders) | 1 (1) | 0 (0)
ELEVATED ALKALINE PHOSPHATASE (Investigations) | 0 (0) | 1 (1)
ELEVATED ALT (Investigations) | 0 (0) | 1 (1)
ELEVATED AST (Investigations) | 0 (0) | 1 (1)
ELEVATED GGT (Investigations) | 0 (0) | 1 (1)
ELEVATED SERUM BILE ACIDS (Investigations) | 0 (0) | 1 (1)
LEFT EAR ERYTHEMA PRESENT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a joint publication is not submitted within 18-24 months after study completion, PI shall have the right to submit to sponsor a proposed results communication based on results at their institution. Sponsor can review proposed results communications prior to public release, can request removal of confidential information, and can embargo communications regarding trial results for up to 105-120 days after submission to sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT03394781/Prot_SAP_000.pdf